CLINICAL TRIAL: NCT05001516
Title: A Phase I, First-in-Human, Open-Label, Dose Escalation and Expansion Study of TPX4589 in Patients With Claudin(CLDN)18.2-Positive Advanced Solid Tumors
Brief Title: Study of Turning Point Therapeutics LM-302 in Patients With Advance Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Turning Point Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA128-1033; CA128-1033 (Other: BMS Protocol ID); LM-302 (TPX4589) (Other: Turning Point Therapeutics Protocol ID)
Record Dates: First submitted 2021-07-27; First posted 2021-08-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Arm1:LM302 0.2 mg/kg i.v., QW×3 weeks group; Arm2:LM302 0.4 mg/kg i.v., QW×3 weeks group; Arm3:LM302 0.8 mg/kg i.v., QW×3 weeks group; Arm4:LM302 1.6 mg/kg i.v., QW×3 weeks group; Arm5:LM302 2.4 mg/kg i.v., QW×3 weeks group; Arm6:LM302 2.8 mg/kg i.v., QW×3 weeks group;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LM302 Dose Escalation Level 1, 0.2 mg/kilogram(kg), (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  first dose: 0.2mg/kg i.v. every 3 weeks (1 cycle=21 days) , n=1;
  Interventions: Drug: LM-302
- LM302 Dose Escalation Level 2, 0.4 mg/kg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  second dose: 0.4mg/kg i.v. every 3 weeks (1 cycle=21 days) , n=3;
  Interventions: Drug: LM-302
- LM302 Dose Escalation Level 3, 0.8 mg/kg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  third dose: 0.8mg/kg i.v. every 3 weeks (1 cycle=21 days) , n=6;
  Interventions: Drug: LM-302
- LM302 Dose Escalation Level 4, 1.6mg/kg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  fourth dose: 1.6mg/kg i.v. every 3 weeks (1 cycle=21 days) , n=6;
  Interventions: Drug: LM-302
- LM302 Dose Escalation Level 5, 2.4mg/kg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  fifth dose: 1.6mg/kg i.v. every 3 weeks (1 cycle=21 days) , n=9;
  Interventions: Drug: LM-302
- LM302 Dose Escalation Level 6, 2.8mg/kg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  sixth dose: 1.6mg/kg i.v. every 3 weeks (1 cycle=21 days) , n=12;
  Interventions: Drug: LM-302

INTERVENTIONS:
Drug: LM-302 — All subjects will be administered every 3 weeks (1 cycle=21 days) with a dose of LM-302 intravenous infusion on day 1 until meet the criteria of treatment discontinuation or withdraw, whichever occurs earlier.

SUMMARY:
A Phase I, First-in-Human, Open-Label, Dose Escalation and Expansion Study of LM-302 in Patients with CLDN18.2-Positive Advanced Solid Tumors

DETAILED DESCRIPTION:
A Phase I, First-in-Human, Open-Label, Dose Escalation and Expansion Study of LM-302 in Patients with CLDN18.2-Positive Advanced Solid Tumors

The study schedule includes screening visit (28 days prior to accept the investigational medicinal product (IMP)), treatment visit (accept IMP for the first time to the end of treatment (EOT)/early withdrawal), and follow-up visit (28 days after the EOT/early withdrawal).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are fully informed of the purpose, nature, method and possible adverse reactions of the study, and are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure;
* Aged ≥18 years old when sign the ICF, male or female;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, and no deterioration within 2 weeks prior to the first dose;
* Life expectancy ≥ 3 months;
* Phase Ⅰa (Dose Escalation): Subjects must have histological or cytological confirmation of recurrent or refractory advanced solid tumors, and have progressed on standard therapy, or are intolerable for available standard therapy , or there is no available standard therapy. The advanced solid tumors include but not limit to gastric and gastroesophageal junction adenocarcinoma, esophageal adenocarcinoma, pancreatic carcinoma, biliary tract carcinoma, colorectal carcinoma, ovarian carcinoma.
* Claudin18.2(CLDN18.2) status will be tested by central immunohistochemistry (IHC) testing for the enrolled subjects if the archived tumor tissue samples are available, and the enrolment is not dependent on the CLDN18.2's status.
* CLDN18.2 positive may be required for the high dose levels as determined by Safety Monitoring Committee(SMC), the subjects need to have CLDN 18.2 positive available before enrolled and dosed, and the tumor types are limited to the types listed as phase Ib (Dose expansion).
* Phase Ib (Dose Expansion): Subjects must have histological or cytological confirmation of recurrent or refractory CLDN18.2 positive* advanced solid tumors, and have progressed on standard therapy, or are intolerable for available standard therapy , or there is no available standard therapy. The advanced solid tumors include the following or the specific tumor types that are determined by SMC:
* Gastric and gastroesophageal junction adenocarcinoma;
* Pancreatic carcinoma;
* Biliary tract carcinoma;
* Colorectal carcinoma with known Microsatellite instability-high(MSI-H)/Different Mismatch Repair(dMMR);
* Esophageal adenocarcinoma;
* Ovarian mucinous carcinoma;

  *CLDN18.2-positive: defined as CLDN18.2 expression confirmed by central immunohistochemistry (IHC) test and with a staining intensity of 1+ to 3+ in ≥ 10% of the tumor cell. At least 3 subjects with a staining intensity of 2+ to 3+ in ≥ 40% of the tumor cells should be included for the dose expansion stage.
* At least one evaluable lesion (including measurable and unmeasurable) for phase Ia dose escalation, and one measurable lesion for phase Ib dose expansion, according to RECIST v1.1;
* Subjects must show appropriate organ and marrow function in laboratory examinations within 7 days prior to the first dose:
* Bone marrow reserve: Platelet count (PLT) ≥ 90 × 109/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Haemoglobin ≥ 9 g/dL, without receiving Erythropoietin(EPO), G-Colony-Stimulating Factor(CSF), or Granulocyte-Macrophage Colony Stimulating Factor(GM-CSF) within 14 days and blood transfusion including red blood cell and platelet transfusion in at least 7 days prior to first dose;
* Coagulation function: International Normalized Ratio(INR) ≤ 1.5; Activated Partial Thromboplastin Time(APTT) ≤ 1.5 × ULN;
* Liver function: Total bilirubin ≤ 1.5 × ULN (Subjects with Gilbert's Syndrome are allowed if total bilirubin ≤ 3 × ULN); Aspartate Transaminase(AST) and Alanine Aminotransferase(ALT) ≤ 2.5 × ULN without liver metastases (≤ 5 × ULN if liver metastases are present); Albumin ≥ 2.5 g/dL;
* Kidney function: Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min (using Cockcroft-Gault formula);
* Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%; QT interval (QTcF) ≤ 480 ms;
* Subjects who are able to communicate we

Exclusion Criteria:

* Exposure to any IMP, or participate in any other clinical trial within 21 days prior to 1st dosing of LM-302;
* Subjects with anti-tumor treatment within 21 days prior to 1st dosing of LM-302, including radiotherapy, chemotherapy, biotherapy, endocrine therapy and immunotherapy, etc. Following treatments have different time limits:
* Local small-scale palliative radiotherapy (bone metastasis radiotherapy to control pain) within 14 days prior to 1st dosing;
* Oral anti-tumor therapy, including fluorouracil antitumor drugs and small molecular targeted drugs, etc. within 14 days or 5 half-life of the drug (whichever is shorter) prior to 1st dosing;
* Traditional Chinese medicine with anti-tumor indication within 14 days prior to 1st dosing.
* Nitrosourea or Mitomycin C within 42 days prior to 1st dosing.
* Any adverse event from prior anti-tumor therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0 (Except for toxicities without safety risk judged by the investigator, such as alopecia, and other ≤ grade 2 long term toxicities);
* Pre-existing peripheral sensory or motor neuropathy ≥ Grade 2;
* Subjects with uncontrolled tumor-related pain. Subjects requiring analgesic treatment must be on a stable regimen before participating in the study. Symptomatic lesions amenable by palliative radiotherapy (e.g., bone metastases or metastases causing nerve damage) should be treated prior to enrolment. For the asymptomatic metastatic lesions whose further growth would likely cause functional defects or intractable pain, if appropriate, local treatment should be considered before enrolment;
* Subjects with known central nervous system (CNS) or meningeal metastasis;
* Subjects who have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures;
* Subjects who are allergic or hypersensitive to LM-302 (The excipients are L-Glutamic acid, L-Arginine, Trehalose dihydrate and polysorbate 80 (for injection)) or similar products;
* Subjects who have received the treatment targeting to CLDN18.2 or Monomethyl Auristatin E(MMAE) based Antibody-Drug Conjugates (ADCs):
* Subjects who have received the treatment with ADCs targeting to CLDN18.2 are not eligible;
* Subjects who were intolerable to the treatment with MMAE based ADCs or anti-CLDN18.2 antibodies are not eligible, but can be enrolled if they were tolerable to the treatments and have experienced a 28-day's washout period prior to 1st dosing of LM-302;
* For Phase Ib (Dose Expansion), subjects who were not response to the treatment with MMAE based ADCs or anti-CLDN18.2 antibodies are not eligible;
* Administrate strong inhibitors/strong inducers of CYP3A4 within 14 days prior to 1st dosing of LM-302;
* Subjects with known active keratitis or corneal ulcerations. Subjects with superficial punctate keratitis are allowed if the disorder is being adequately treated in the opinion of the investigator.
* Use of any live vaccines (e.g., against infectious diseases such as influenza, varicella, COVID-19, etc.) within 28 days prior to 1st dosing of LM-302;
* Subjects with the history of interstitial lung disease or drug-induced interstitial lung disease/pneumonitis;
* Subjects who are taking therapeutic doses of anticoagulants such as heparin or vitamin K antagonists (except for preventive treatment at a stable dose);
* Subjects with gastric outlet obstruction, persistent recurrent vomiting or uncontrolled/severe gastrointestinal hemorrhage, or ulcer within 28 days prior to 1st dosing of LM-302;
* Subjects who received major surgery or interventional treatment within 28 days prior to 1st dosing of LM-302 (excluding tumor biopsy, puncture, etc.);
* Subjects who have other active malignancies which are likely to require the treatment;
* Subjects who have severe cardiovascular disease, including but not limited to:
* Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, and II-III degree atrioventricular block, etc.;
* Thromboembolic events requiring therapeutic anticoagulation, or equipped with venous filters;
* Cardiac insufficiency of grade III~IV according to the New York Heart Association (NYHA) standards;
* Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other cardiovascular and cerebrovascular events of grade 3 or above occurred within 6 months prior to 1st dosing of LM-302;
* Clinically uncontrollable hypertension;
* Subjects who have uncontrolled or severe illness, including but not limited to ongoing or active infection (e.g., active Corona Virus Disease 2019（COVID-19）/Severe Acute Respiratory Syndromes(SARS)-COVID-2 infection, etc.) requiring antibiotics and/or other therapeutic administration, while SARS-COVID-2 testing is not mandatory for study entry, and the testing should follow local clinical practice guidelines/standards.
* Subjects who have a history of immunodeficiency disease, including other acquired or congenital immunodeficiency diseases, or organ transplantation, or allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation;
* HIV infection, active Hepatitis B Virus(HBV) and Hepatitis C Virus(HCV)infection, with the exception:
* Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-hepatitis B core(HBc)] and absence of HBsAg), as well as with normal liver function are eligible. Otherwise, if HBV infection was indicated, those with HBV DNA < 500 IU/ML (or equivalent level) and normal liver function, combined with clinical manifestations, judged by the investigator to exclude active infection can be enrolled;
* Subjects with positive HCV antibody but negative hepatitis C virus RNA test results and normal liver function are eligible.
* Child-bearing potential female who have positive results in pregnancy test or are lactating;
* Subjects who have psychiatric illness or disorders that may preclude study compliance;
* Subject who is judged as not eligible to participate in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Cycle 1 of each cohort. Duration of one cycle is 21 days
  DLT is defined as a toxicity (adverse event at least possibly related to LM302) occurring during the DLT observation period
Number of participants with adverse events and serious adverse events | From the first administration in Cycle 1 date 1(C1D1)up to 1 year
  The safety profile of LM302 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Change in Vital Signs-ear temperature | Baseline C1D1through approximately 1 year after first administration of LM302
  Change in vital signs-ear temperature will be measured after the subject has been fully rested
Change in Vital Signs-pulse rate | Baseline C1D1through approximately 1 year after first administration of LM302
  Change in vital signs-pluse rate will be measured after the subject has been fully rested.
Change in Vital Signs-systolic pressure | Baseline C1D1through approximately 1 year after first administration of LM302
  Change in vital signs-systolic pressure will be measured after the subject has been fully rested.
Change in Vital Signs-diastolic blood pressure | Baseline C1D1through approximately 1 year after first administration of LM302
  Change in vital signs-diastolic blood pressure will be measured after the subject has been fully rested.
Change in Physical examination-weight | Baseline C1D1through approximately 1 year after first administration of LM302
  Change in Physical examination-weight will be measured with only light clothes
Incidence of Abnormal Clinical Laboratory Test Results-hematology | Baseline C1D1through approximately 1 year after first administration of LM302
  Number of participants with incidence of abnormal clinical lab test results like hematology will be assessed.
Incidence of Abnormal Clinical Laboratory Test Results-Biochemistry | Baseline C1D1through approximately 1 year after first administration of LM302
  Number of participants with incidence of abnormal clinical lab test results like Biochemistry will be assessed
Incidence of Abnormal Clinical Laboratory Test Results-Urinalysis | Baseline C1D1through approximately 1 year after first administration of LM302
  Number of participants with incidence of abnormal clinical lab test results like Urinalysis will be assessed.
Incidence of Abnormal Clinical Laboratory Test Results-Coagulation test | Baseline C1D1through approximately 1 year after first administration of LM302
  Number of participants with incidence of abnormal clinical lab test results like Coagulation test will be assessed
Change in Electrocardiogram (ECG)-(R wave)RR interval | Baseline C1D1through approximately 1 year after first administration of LM302
  RR interval of 12-lead ECG will be performed in the supine position after the patients are fully rested at each timepoint for once. RR is the standard heart rate which calculated by 60 divided by heart rate.
Change in Electrocardiogram (ECG)-QT interval | Baseline C1D1through approximately 1 year after first administration of LM302
  QT interval of 12-lead ECG will be performed in the supine position after the patients are fully rested at each timepoint for once.
Change in Electrocardiogram (ECG)-QRS duration | Baseline C1D1through approximately 1 year after first administration of LM302
  QRS duration of 12-lead ECG will be performed in the supine position after the patients are fully rested at each timepoint for once.

SECONDARY OUTCOMES:
Area under the serum concentration versus time curve within one dosing interval (AUCtau) | Up to 1 year
  Blood samples will be collected at time points of 0 h, immediately after infusion stop, as well as at 1 h,4 h, 8 h, 24 h, 48 h (Day 3), 168 h (Day 8), and 336 h (Day 15) after infusion stop in cycle 1 and cycle 4; 0 h in cycle 2, cycle 3 and cycle 5; pre-dose (0 h) will be collected in every other cycle for the subsequent cycles. i.e., in cycle 6, cycle 8, … etc.; at EOT/early withdraw from the study (if the EOT/early withdraw occur when PK blood sampling isn't stipulated). The timepoints of PK sample may be adjusted base on the human PK data. The blood samples for PK analysis will be collected as much as possible if the subjects end of treatment/early withdraw.
Volume of distribution at steady state (Vss) | Up to 1 year
  To determine the pharmacokinetics (PK) profile of LM302
Maximum serum concentration (Cmax) | Up to 1 year
  To determine the pharmacokinetics (PK) profile of LM302
Minimum serum concentration（Cmin） | Up to 1 year
  To determine the pharmacokinetics (PK) profile of LM302
Time to reach maximum serum concentration (Tmax) | Up to 1 year
  To determine the pharmacokinetics (PK) profile of LM302
Clearance (CL) | Up to 1 year
  To determine the pharmacokinetics (PK) profile of LM302
Terminal half-life (T1/2) | Up to 1 year
  To determine the pharmacokinetics (PK) profile of LM302
Dose proportionality | Up to 1 year
  To determine the pharmacokinetics (PK) profile of LM302
Objective response rate of LM-302. | Up to 1 year
  Preliminary anti-tumor activity of LM-302 according to RECIST v1.1 assessed by investigator: objective response rate (ORR, complete response(CR)+ partial response(PR))
Duration of response of LM-302. | Up to 1 year
  Preliminary anti-tumor activity of LM-302 according to RECIST v1.1 assessed by investigator: Duration of response (DOR)
Disease control rate of LM-302. | Up to 1 year
  Preliminary anti-tumor activity of LM-302 according to RECIST v1.1 assessed by investigator: disease control rate (DCR, CR+PR+SD)
Progression-free survival of LM-302. | Up to 1 year
  Preliminary anti-tumor activity of LM-302 according to RECIST v1.1 assessed by investigator:progression-free survival (PFS)
To assess the immunogenicity of LM-302; | Up to 1 year
  Blood samples collected for Anti-Drug Antibody(ADA) assessment will be performed at 0 h of Day 1 (within 30 min prior to infusion) in cycle 1 to Cycle 5; 0 h of Day 1 in every other cycle (within 30 min prior to infusion) for the subsequent cycles, i.e., in cycle 6, cycle 8, … etc., the EOT/early withdraw from the study and safety follow-up. Nab will be detected if necessary.

OTHER OUTCOMES:
To explore the correlation between CLDN18.2 expression and anti-tumor activity of LM-302 | Up to 2 years
  Test CLDN18.2 expression and anti-tumor activity of LM-302

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - Local Institution - 0013, Duarte, California
  - Local Institution - 0017, Fullerton, California
  - Local Institution - 0012, Lafayette, Indiana
  - Local Institution - 0020, Paramus, New Jersey
  - Local Institution - 0018, New York, New York
  - Local Institution - 0016, Oklahoma City, Oklahoma
  - Local Institution - 0015, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com